CLINICAL TRIAL: NCT01927068
Title: Prospective, Single-Arm, Global Multi-Center Study to Evaluate Treatment of Obstructive Superficial Femoral Artery (SFA) and/or Popliteal Lesions With a Novel Paclitaxel-Coated Percutaneous Angioplasty (PTA) Balloon and in In-Stent Restenosis
Brief Title: STELLAREX: ILLUMENATE Global and In-Stent Restenosis (ISR)
Acronym: ILLUMENATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spectranetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-1005; CP-1005B (Other: Spectranetics)
Record Dates: First submitted 2013-07-25; First posted 2013-08-22 (Estimated); Results first posted 2022-03-15 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Global Cohort 1 (Experimental): All subjects to be treated with the Stellarex 035 Drug Coated Balloon (DCB) for Percutaneous Transluminal Angioplasty (PTA).The drug coating is paclitaxel (PTX).
  Interventions: Device: Stellarex 0.035" Over-the-Wire (OTW) drug-coated angioplasty balloon (Stellarex DCB)
- ISR Cohort 2 (Experimental): All subjects to be treated with the Stellarex 035 Drug Coated Balloon (DCB) for Percutaneous Transluminal Angioplasty (PTA).The drug coating is paclitaxel (PTX).
  Interventions: Device: Stellarex 0.035" Over-the-Wire (OTW) drug-coated angioplasty balloon (Stellarex DCB)

INTERVENTIONS:
Device: Stellarex 0.035" Over-the-Wire (OTW) drug-coated angioplasty balloon (Stellarex DCB) — Percutaneous Transluminal Angioplasty will be completed using a 2.0 micrograms per square millimeter. Paclitaxel-Coated Balloon. Balloon will be inflated to a size appropriate for the target vessel, as determined by the physician. Total balloon inflation time is determined by the physician, but no less than one minute.
  Other Names: CVI Paclitaxel-Coated PTA Balloon Catheter

SUMMARY:
Cohort 1: Single-Arm, multicenter study to continue to assess the safety and performance of the Stellarex 035 Drug Coated Balloon (formerly known as the Cardiovascular Ingenuity (CVI) Paclitaxel-Coated PTA Balloon Catheter) in the treatment of de novo or restenotic lesions in the superficial femoral and/or popliteal arteries.

Cohort 2: To evaluate this patient population for treatment of in-stent restenotic lesions.

DETAILED DESCRIPTION:
Cohort 1:

The purpose of this single arm study is to continue to assess safety and performance of the Stellarex 035 DCB in the treatment of de novo or restenotic lesions in the superficial femoral (SFA) and/or popliteal arteries.

Cohort 2:

A second cohort is being added to evaluate this patient population for treatment of in-stent restenotic lesions.

Cohort 1:

Prospective, multi-center, single-arm study.

Cohort 2:

Prospective, multi-center, single-arm study compared to a historical control.

Cohort 1:

Follow-up assessments will occur at discharge, 1 month, 6 months, 12 months, 24 months, 36 months, 48 months, and 60 months following the study procedure.

Cohort 2:

Follow-up assessments will occur at discharge, 1 month, 6 months, 12 months, 24 months and 36 months following the study procedure.

ELIGIBILITY:
Cohort 1: General Inclusion Criteria:

1. Has symptomatic leg ischemia, requiring treatment of the SFA and/or popliteal artery.
2. Has a Rutherford Clinical Category of 2 - 4. Note: Rutherford Clinical Category 2 subjects should be entered into the study if conservative treatment has been unsuccessful.
3. Is ≥18 years old.
4. Has life expectancy >1 year.
5. Is able and willing to provide written informed consent prior to study specific procedures.
6. Is willing and capable of complying with the required follow-up visits, testing schedule and medication regimen.

Cohort 1: Angiographic Inclusion Criteria:

1. Has evidence at the target lesion(s) of clinically and hemodynamically significant de novo stenosis or restenosis, or occlusion, in the SFA (1 cm distal to the ostium of the profunda) and/or popliteal artery (proximal to the popliteal trifurcation), confirmed by angiography.
2. Has target limb with at least one patent (<50% stenosis) tibio-peroneal run-off vessel to the foot confirmed by baseline angiography or magnetic resonance angiography (MRA) or computed tomography angiography (CTA). Note: Treatment of outflow disease is NOT permitted.
3. Has 1 or 2 target lesion(s) with a cumulative lesion(s) length of no more than 20 cm. Note: A maximum of two (2) lesions can be treated if the cumulative total lesion length (i.e. the combined length of both lesions) is less than or equal to 20cm.
4. Has target lesion(s) located >2 cm from any stent if the target vessel was previously stented.
5. Has a reference vessel diameter of 4 - 6 mm by visual estimate.
6. Has a successful exchangeable guidewire crossing of the lesion(s).

Cohort 1: General Exclusion Criteria:

1. A female who is pregnant, of childbearing potential not taking adequate contraceptive measures, or nursing; or a male intending to father children during the study.
2. Has significant gastrointestinal bleeding or any coagulopathy that would contraindicate the use of anti-platelet therapy
3. Has known intolerance to study medications, paclitaxel or contrast agents that in the opinion of the investigator cannot be adequately pre-treated.
4. Is currently participating in another investigational device or drug study that would interfere with study endpoints.
5. Has history of hemorrhagic stroke within 3 months.
6. Has surgical or endovascular procedure of the target limb within 14 days prior to the index procedure.
7. Has any planned surgical intervention (requiring hospitalization) or endovascular procedure within 30 days after the index procedure.
8. Has had a previous peripheral bypass affecting the target limb.
9. Has unstable angina pectoris, myocardial infarction, liver failure, renal failure or chronic kidney disease (dialysis dependent, or serum creatinine ≥2.5 mg/dL) within 30 days of the index procedure.

Cohort 1: Angiographic Exclusion Criteria:

1. Has significant stenosis (≥50%) or occlusion of inflow tract that is not successfully revascularized (<30% residual stenosis without death or major vascular complication) prior to treatment of the target lesion(s). Only treatment of target lesion(s) is acceptable after successful treatment of inflow iliac artery lesion(s).
2. Has an acute or sub-acute intraluminal thrombus within the target vessel.
3. Has in-stent restenosis or restenosis of the target lesion following previous treatment with a drug-coated balloon.
4. Has an aneurysm (at least twice the reference vessel diameter) located in the target vessel, abdominal aorta, iliac, or popliteal arteries.
5. Has perforation, dissection or other injury of the access or target vessel requiring stenting or surgical intervention prior to enrollment.
6. Has no normal arterial segment proximal to the target lesion in which duplex ultrasound velocity ratios can be measured.
7. Requires use of adjunctive therapies (i.e., laser, atherectomy, cryoplasty, scoring/cutting balloons, brachytherapy).
8. Has severe calcification that precludes adequate PTA treatment.

Cohort 2: General Inclusion Criteria:

1. Has symptomatic leg ischemia, requiring treatment of the SFA and/or popliteal artery.
2. Has a Rutherford Clinical Category of 2 - 4. Note: Rutherford Clinical Category 2 subjects should be entered into the study if conservative treatment has been unsuccessful.
3. Is between 18-85 years old.
4. Has life expectancy >1 year.
5. Is able and willing to provide written informed consent prior to study specific procedures.
6. Is willing and capable of complying with the required follow-up visits, testing schedule and medication regimen.
7. History of previous femoropopliteal nitinol stenting which is suspect for in-stent restenosis.
8. The patient has a resting ankle-brachial index (ABI) <0.9 or an abnormal exercise ABI (<0.9) if resting ABI is normal. Patient with incompressible arteries (ABI>1.2) must have a toe-brachial index (TBI) <0.7 in target limb.

Cohort 2: Angiographic Inclusion Criteria:

1. Has angiographic evidence of significant restenosis (≥50% by visual estimate) within a previously deployed femoropopliteal bare nitinol stent(s) including ISR Class I, II or III.
2. Has target limb with at least one patent (<50% stenosis) tibio-peroneal run-off vessel to the foot confirmed by baseline angiography or magnetic resonance angiography (MRA) or computed tomography angiography (CTA). Note: Treatment of outflow disease is NOT permitted.
3. Total target treatment length of in-stent restenosis must be ≥4.0 cm in length and may include a single lesion or a multifocal lesion within the femoropopliteal segment (This includes the proximal, mid, and/or distal SFA and PI, P2 and/or P3 segment of the popliteal artery). Edge restenosis may be treated provided the lesion extends no more than 3 cm outside the margin of the stent (proximal and/or distal margin).
4. Has target lesion(s) located >2 cm from any stent if the target vessel was previously stented.
5. Has a reference vessel diameter of 4 - 6 mm by visual estimate.
6. Has a successful exchangeable guidewire crossing of the lesion(s).

Cohort 2: General Exclusion Criteria:

1. A female who is pregnant, of childbearing potential not taking adequate contraceptive measures, or nursing; or a male intending to father children during the study.
2. Has significant gastrointestinal bleeding or any coagulopathy that would contraindicate the use of anti-platelet therapy.
3. Has known intolerance to study medications, paclitaxel or contrast agents that in the opinion of the investigator cannot be adequately pre-treated.
4. Is currently participating in another investigational device or drug study that would interfere with study endpoints.
5. Has history of hemorrhagic stroke within 3 months including those within <60 days with an unresolved walking impairment.
6. Has surgical or endovascular procedure of the target limb within 3 months prior to the index procedure.
7. Has any planned surgical intervention (requiring hospitalization) or endovascular procedure within 30 days after the index procedure.
8. Has had a previous peripheral bypass affecting the target limb.
9. Has unstable angina pectoris, myocardial infarction within 60 days, liver failure, renal failure or chronic kidney disease (dialysis dependent, or serum creatinine ≥2.5 mg/dL) within 30 days of the index procedure.
10. History of previous femoropopliteal stenting in the target lesion with drug eluting stents or covered stents (endografts).

Cohort 2: Angiographic Exclusion Criteria:

1. Ipsilateral and/or contralateral iliac (or common femoral) artery stenosis

   ≥50% diameter stenosis (DS) that is not successfully treated prior to index procedure (e.g. where a perforation occurred requiring a covered stent) or with final residual stenosis ≥ 30% documented by angiography.
2. Identification of any lesion of the native vessel (excludes ISR) above the target stent in the femoropopliteal segment >50% that is not successfully treated prior to index procedure (e.g. complication requiring additional treatment) or with final residual stenosis >30% documented by angiography. Drug eluting stent (DES) and drug coated balloon (DCB) will not be allowed. The lesion length must be treatable with a single stent (if required). The lesion must not be contiguous with the target lesion; at least 2 cm of normal appearing vessel between the lesion and target lesion/ target stent or between deployed stent (if required) and the target lesion/ target stent.
3. Has an acute or sub-acute intraluminal thrombus within the target vessel.
4. Has an aneurysm (at least twice the reference vessel diameter) located in the target vessel, abdominal aorta, iliac, or popliteal arteries.
5. Has perforation, dissection or other injury of the access or target vessel requiring stenting or surgical intervention prior to enrollment.
6. Has no normal arterial segment proximal to the target lesion in which duplex ultrasound velocity ratios can be measured.
7. Requires use of adjunctive therapies (i.e., laser, atherectomy, cryoplasty, scoring/cutting balloons, brachytherapy).
8. Grade 4 or 5 stent fracture affecting target stent or proximal to the target stent, or where evidence of stent protrusion into the lumen is noted on angiography in 2 orthogonal views.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 499 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2022-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zeller, MBChB, FRANZCR, Principal Investigator — Herz-Zentrum Bad Krozingen, Germany; Andrew Holden, MD, Principal Investigator — Auckland Hospital, New Zealand; Yann Goueffic, MD, Principal Investigator — Hopital Nord Laennec, France
Locations (44):
- Australia (6):
  - The Wesley St. Andrew Research Institute Ltd., Auchenflower
  - Flinders Medical Centre, Bedford
  - Royal Brisbane and Women's Hospital, Brisbane
  - Monash Medical Centre at Dandenong Campus, Dandenong
  - The Alfred Hospital, Melbourne
  - Sir Charles Gairdner Hospital, Nedlands
- Medizinische Universität Graz - Univ. Klinik für Innere Medizin, Graz, Austria
- Belgium (8):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - Middelheim Hospital, Antwerp
  - Imelda Hospital, Bonheiden
  - AZ Sint-Blasius, Dendermonde
  - ZOL Campus Sint Jan, Genk
  - Universitair Ziekenhuis Gent, Ghent
  - University Clinic Leuven, Leuven
  - Regionaal Ziekenhuis Heilig Hart Tienen, Campus Mariëndal - MCT, Vascular Surgery Department, Tienen
- France (7):
  - CHU de Clermont-Ferrand, Hôpital Gabriel Montpied, Clermont-Ferrand
  - CHU de Lyon, Hôpital Edouard Herriot, Lyon
  - Hopital de Ia Timone, Marseille
  - CHU de Nantes, Hôpital Nord Laennec, Nantes
  - Hôpital Européen georges Pompidou, Paris
  - CHU de Rennes, Hôpital Pontchaillou, Rennes
  - Clinique Pasteur, Toulouse
- Germany (8):
  - Universitats-Herzzentrum Freiburg - Bad Krozingen, Bad Krozingen
  - Jüdisches Krankenhaus Berlin, Berlin
  - Medizinische Universitätsklinik III, Heidelberg
  - Klinikum Immenstadt, Herz-und Gefässzentrum Oberallgäu-Kempten, Immenstadt im Allgäu
  - SRH Klinikum Karlsbad-Langensteinbach, Langensteinbach
  - University Leipzig Medical Center, Leipzig
  - RoMed Klinikum Rosenheim, Rosenheim
  - Universitatsklinik, Abteilung Für Diagnostische und Inverventionelle Radiologie, Tübingen
- Italy (3):
  - Ospedali Riuniti - SOD, Ancona
  - Villa Maria Eleonora Hospital, Palermo
  - S.C. Chirurgia Vascolare ed Endovascolare, Perugia
- New Zealand (4):
  - Auckland City Hospital, Auckland
  - Middlemore Hospital, Auckland
  - Waikato Hospital, Hamilton
  - Wellington Hospital, Wellington
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Instytut Hematologii i Transfuzjologii, Warsaw
- Spain (2):
  - Centre d'Atencio Integral Hospital Dos de Maig, Barcelona
  - Hospital Universitario Quirón de Madrid, Madrid
- United Kingdom (3):
  - Imperial College Academic and Healthcare NHS Trust, St. Mary's Hospital, London
  - King's College, London
  - UCL Division of Surgery and Interventional Science, London

REFERENCES:
- [Derived] Gray WA, Jaff MR, Parikh SA, Ansel GM, Brodmann M, Krishnan P, Razavi MK, Vermassen F, Zeller T, White R, Ouriel K, Adelman MA, Lyden SP. Mortality Assessment of Paclitaxel-Coated Balloons: Patient-Level Meta-Analysis of the ILLUMENATE Clinical Program at 3 Years. Circulation. 2019 Oct;140(14):1145-1155. doi: 10.1161/CIRCULATIONAHA.119.040518. Epub 2019 Sep 30. PMID 31567024

RESULTS

PARTICIPANT FLOW:
Groups:
- Global Cohort 1: The purpose of this single arm cohort is to continue to assess safety and performance of the Stellarex 035 DCB in the treatment of de novo or restenotic lesions in the superficial femoral (SFA) and/or popliteal arteries.
  All subjects to be treated with the Stellarex 035 Drug Coated Balloon (DCB) for Percutaneous Transluminal Angioplasty (PTA).The drug coating is paclitaxel (PTX).
  Stellarex 0.035" Over-the-Wire (OTW) drug-coated angioplasty balloon (Stellarex DCB): Percutaneous Transluminal Angioplasty will be completed using a 2.0 micrograms per square millimeter. Paclitaxel-Coated Balloon. Balloon will be inflated to a size appropriate for the target vessel, as determined by the physician. Total balloon inflation time is determined by the physician, but no less than one minute.
- ISR Cohort 2: The goal of cohort 2 is to evaluate this patient population for treatment of in-stent restenotic lesions, which is different than the population in cohort 1.
  All subjects to be treated with the Stellarex 035 Drug Coated Balloon (DCB) for Percutaneous Transluminal Angioplasty (PTA).The drug coating is paclitaxel (PTX).
  Stellarex 0.035" Over-the-Wire (OTW) drug-coated angioplasty balloon (Stellarex DCB): Percutaneous Transluminal Angioplasty will be completed using a 2.0 micrograms per square millimeter. Paclitaxel-Coated Balloon. Balloon will be inflated to a size appropriate for the target vessel, as determined by the physician. Total balloon inflation time is determined by the physician, but no less than one minute.
Period: Overall Study
Arm/Group | Global Cohort 1 | ISR Cohort 2
Started | 370 | 129
Completed | 262 | 121
Not Completed | 108 | 8
Not completed — Death | 37 | 3
Not completed — Withdrawal by Subject | 50 | 3
Not completed — Lost to Follow-up | 10 | 2
Not completed — Physician Decision | 9 | 0
Not completed — Missed last follow-up visit | 2 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Participants are based on the Intent-to-Treat (ITT) analysis set meaning all participants enrolled in the study. The outcome measures and safety results for the adverse events section will be based on the modified Intent-to-Treat set (mITT). The mITT is all participants in the ITT set who did not receive a bailout stent. Seven participants received a bailout stent so the mITT is composed of 122 participants.
Groups:
- Global Cohort 1: The purpose of this single arm study is to continue to assess safety and performance of the Stellarex 035 DCB in the treatment of de novo or restenotic lesions in the superficial femoral (SFA) and/or popliteal arteries.
  All subjects to be treated with the Stellarex 035 Drug Coated Balloon (DCB) for Percutaneous Transluminal Angioplasty (PTA).The drug coating is paclitaxel (PTX).
  Stellarex 0.035" Over-the-Wire (OTW) drug-coated angioplasty balloon (Stellarex DCB): Percutaneous Transluminal Angioplasty will be completed using a 2.0 micrograms per square millimeter. Paclitaxel-Coated Balloon. Balloon will be inflated to a size appropriate for the target vessel, as determined by the physician. Total balloon inflation time is determined by the physician, but no less than one minute.
- ISR Cohort 2: Same patient population in Cohort 1, but cohort 2 is to evaluate this patient population for treatment of in-stent restenotic lesions.
  All subjects to be treated with the Stellarex 035 Drug Coated Balloon (DCB) for Percutaneous Transluminal Angioplasty (PTA).The drug coating is paclitaxel (PTX).
  Stellarex 0.035" Over-the-Wire (OTW) drug-coated angioplasty balloon (Stellarex DCB): Percutaneous Transluminal Angioplasty will be completed using a 2.0 micrograms per square millimeter. Paclitaxel-Coated Balloon. Balloon will be inflated to a size appropriate for the target vessel, as determined by the physician. Total balloon inflation time is determined by the physician, but no less than one minute.
- Total: Total of all reporting groups
Arm/Group | Global Cohort 1 | ISR Cohort 2 | Total
Number analyzed (Participants) | 370 | 129 | 499
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (9.3) | 69 (9.4) | NA (NA) — Cohort 1 and cohort 2 are two distinct populations with separate study inclusion/exclusion criteria. The two populations are not poolable. The two cohorts represent different populations with respect to the disease state. A patient with ISR as well as PAD is different than a PAD patient alone. For that reason, we believe that the two populations should remain separate as pooling the overall population does not provide any value to the reader.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 46 | 145
  Male | 271 | 83 | 354
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2 | 1 | 3
  White | 327 | 128 | 455
  Asian | 4 | 0 | 4
  Native Hawaiian or Pacific Islander | 2 | 0 | 2
  Other | 29 | 0 | 29
  Unknown | 6 | 0 | 6
Baseline Ankle-Brachial Index [Mean (Standard Deviation); unit: ratio] — The Ankle-Brachial Index (ABI) is calculated ratio of the highest ankle blood pressure to the highest arm blood pressure. The ABI is a non-invasive tool for screening for Peripheral Artery Disease. Population: The ABI is part of the most missed assessments at baseline which accounts for the missing data. For some participants, ABI is non-measurable or the number too high suggesting non-compressible vessels (with a pressure cuff) and thus cannot be reported.
  ratio
    number analyzed (Participants) | 346 | 118 | 464
    (all) | 0.70 (0.20) | 0.66 (0.18) | NA (NA) — Cohort 1 and cohort 2 are two distinct populations with separate study inclusion/exclusion criteria. The two populations are not poolable. The two cohorts represent different populations with respect to the disease state. A patient with ISR as well as PAD is different than a PAD patient alone. For that reason, we believe that the two populations should remain separate as pooling the overall population does not provide any value to the reader.
Baseline Rutherford-Becker Clinical Category [Count of Participants; unit: Participants] — The Rutherford-Becker Clinical Categories (RCC) are a classification system of chronic limb ischemia ranging from 0 (asymptomatic; no hemodynamically significant occlusive disease) to 6 (major tissue loss, extending above transmetatarsal level, functional foot no longer salvageable). Lower categories represent better clinical status.
  Participants
    RCC 1 | 1 | 0 | 1
    RCC 2 | 124 | 33 | 157
    RCC 3 | 213 | 86 | 299
    RCC 4 | 23 | 9 | 32
    RCC 5 | 9 | 1 | 10
Peripheral Vascular Disease [Count of Participants; unit: Participants] | 295 | 127 | 422
Hypertension [Count of Participants; unit: Participants] | 294 | 102 | 396
Hyperlipidemia [Count of Participants; unit: Participants] | 276 | 101 | 377
Coronary Heart Disease [Count of Participants; unit: Participants]
  Myocardial Infarction | 64 | 21 | 85
  Angina Pectoris | 49 | 10 | 59
  Congestive Heart Failure | 14 | 11 | 25
Previous Percutaneous or Surgical Coronary Revascularization [Count of Participants; unit: Participants] | 123 | 35 | 158
Renal Insufficency [Count of Participants; unit: Participants] | 26 | 20 | 46
Liver Disease [Count of Participants; unit: Participants] | 12 | 6 | 18
Cerebrovascular Disease [Count of Participants; unit: Participants] | 63 | 25 | 88
Chronic Obstructive Pulmonary Disease (COPD) [Count of Participants; unit: Participants] | 49 | 16 | 65
Deep Vein Trhombosis [Count of Participants; unit: Participants] | 8 | 2 | 10
Diabetes [Count of Participants; unit: Participants]
  Type I | 5 | 0 | 5
  Type II | 119 | 49 | 168
Smoker [Count of Participants; unit: Participants]
  Never Smoked | 66 | 23 | 89
  Previous or Current Smoker | 304 | 106 | 410

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Freedom From Device and Procedure-related Death and Freedom From Target Limb Major Amputation and Clinically-driven Target Lesion Revascularization
Description: Freedom from device and procedure-related death through 30 days post-procedure and freedom from target limb major amputation and clinically-driven target lesion revascularization (TLR) through 12 months post-procedure.
Time Frame: Through 12 months post-procedure.
Population: The Modified Intention-to-Treat (mITT) will be comprised of all subjects in the ITT population who do not receive a bailout stent and did not receive provisional treatment for >50% residual stenosis post all assigned treatment or bailout stenting. The primary analysis for both safety and efficacy will be based on the mITT population. In cohort 2, seven patients had bail-out stenting.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Global ISR Cohort 2: The goal of cohort 2 is to evaluate this patient population for treatment of in-stent restenotic lesions, which is different than the population in cohort 1.
  All subjects to be treated with the Stellarex 035 Drug Coated Balloon (DCB) for Percutaneous Transluminal Angioplasty (PTA).The drug coating is paclitaxel (PTX).
  Stellarex 0.035" Over-the-Wire (OTW) drug-coated angioplasty balloon (Stellarex DCB): Percutaneous Transluminal Angioplasty will be completed using a 2.0 micrograms per square millimeter. Paclitaxel-Coated Balloon. Balloon will be inflated to a size appropriate for the target vessel, as determined by the physician. Total balloon inflation time is determined by the physician, but no less than one minute.
Arm/Group | Global Cohort 1 | Global ISR Cohort 2
Number analyzed (Participants) | 370 | 122
percentage of participants | 94.8 [91.9 to 96.6] | 84.1 [77.28 to 90.88]

2. Primary Outcome: Percentage of Lesions Free From Restenosis
Description: Primary patency at 12 months post-procedure. Primary patency is defined as the absence of target lesion restenosis per duplex ultrasound (peak systolic velocity ratio (PSVR) ≤ 2.5) and freedom from clinically-driven target lesion revascularization.
Time Frame: 12 months post-procedure.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Global Cohort 1 | Global ISR Cohort 2
Number analyzed (Participants) | 370 | 122
Number analyzed (Lesions) | 416 | 122
percentage of lesions | 77.8 [73.2 to 81.9] | 58.8 [49.21 to 68.43]

3. Secondary Outcome: Secondary Efficacy Endpoint
Description: The secondary efficacy outcome was freedom from target lesions revascularization (TLR) at 12 months post-procedure and compared to a performance goal.
Time Frame: 12 months post-procedure
Population: The Modified Intention to-Treat (mITT) will be comprised of all subjects in the ITT population who do not receive a bailout stent and did not receive provisional treatment for >50% residual stenosis post all assigned treatment or bailout stenting The primary analysis for safety and efficacy will be based on the mITT population In cohort 2, seven patients had bail-out stenting Data were only collected from Cohort 2 All data for prespecified Primary & Secondary Outcome Measures should be reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Global ISR Cohort 2: The goal of cohort 2 is to evaluate this patient population for treatment of in-stent restenotic lesions, which is different than the population in cohort 1. Data were only collected from Cohort 2. All data for pre-specified Primary and Secondary Outcome Measures should be reported.
  All subjects to be treated with the Stellarex 035 Drug Coated Balloon (DCB) for Percutaneous Transluminal Angioplasty (PTA).The drug coating is paclitaxel (PTX).
  Stellarex 0.035" Over-the-Wire (OTW) drug-coated angioplasty balloon (Stellarex DCB): Percutaneous Transluminal Angioplasty will be completed using a 2.0 micrograms per square millimeter. Paclitaxel-Coated Balloon. Balloon will be inflated to a size appropriate for the target vessel, as determined by the physician. Total balloon inflation time is determined by the physician, but no less than one minute.
Arm/Group | Global ISR Cohort 2
Number analyzed (Participants) | 122
percentage of participants | 83.5 [75.4 to 89.7]

ADVERSE EVENTS:
Time Frame: For cohort 1, the adverse event data reflects 60 months of follow-up post-procedure. For cohort 2, the adverse event data is through 12-months follow-up post-procedure,
Arm/Group | Global Cohort 1 | Global ISR Cohort 2
All-Cause Mortality (participants affected / at risk) | 37/370 | 3/122
Serious Adverse Events (participants affected / at risk) | 291/370 | 65/122
Other Adverse Events (participants affected / at risk) | 343/370 | 93/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Global Cohort 1 (N=370) | Global ISR Cohort 2 (N=122)
Acute Myocardial Infarction (Cardiac disorders) | 17 (18) | 1 (1)
CATHETER SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 12 (12) | 0 (0)
AUTOIMMUNE HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 7 (13) | 0 (0)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 2 (2) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 12 (13) | 1 (1)
ANGINA UNSTABLE (Cardiac disorders) | 7 (9) | 0 (0)
AORTIC VALVE STENOSIS (Cardiac disorders) | 5 (5) | 0 (0)
ARRHYTHMIA (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 8 (9) | 1 (1)
ATRIAL FLUTTER (Cardiac disorders) | 4 (13) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 2 (2) | 0 (0)
CARDIAC DISORDER (Cardiac disorders) | 1 | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 10 (16) | 1 (1)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 (1) | 0 (0)
CARDIOGENIC SHOCK (Cardiac disorders) | 1 (1) | 0 (0)
COR PULMONALE ACUTE (Cardiac disorders) | 1 (1) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 17 (20) | 4 (4)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 3 (4) | 0 (0)
DIASTOLIC DYSFUNCTION (Cardiac disorders) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 4 (4) | 1 (1)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 2 (2) | 0 (0)
PALPITATIONS (Cardiac disorders) | 2 (2) | 0 (0)
SICK SINUS SYNDROME (Cardiac disorders) | 1 (1) | 0 (0)
STRESS CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
TACHYARRHYTHMIA (Cardiac disorders) | 1 (1) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 4 (4) | 0 (0)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 2 (2) | 0 (0)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 3 (3) | 0 (0)
CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1)
DEAFNESS (Ear and labyrinth disorders) | 1 (1) | 0 (0)
MENIERE'S DISEASE (Ear and labyrinth disorders) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0)
GOITRE (Endocrine disorders) | 1 (1) | 0 (0)
HYPERPARATHYROIDISM (Endocrine disorders) | 1 (1) | 0 (0)
CORNEAL DECOMPENSATION (Eye disorders) | 1 (1) | 0 (0)
ECTROPION (Eye disorders) | 1 (1) | 0 (0)
ENTROPION (Eye disorders) | 1 (1) | 0 (0)
EYE HAEMORRHAGE (Eye disorders) | 1 (1) | 0 (0)
LAGOPHTHALMOS (Eye disorders) | 1 (1) | 0 (0)
MACULAR FIBROSIS (Eye disorders) | 1 (1) | 0 (0)
EYELID PTOSIS (Eye disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (4) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0)
BARRETT'S OESOPHAGUS (Gastrointestinal disorders) | 2 (2) | 1 (1)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 (1) | 0 (0)
DENTAL CARIES (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 0 (0)
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 1 (1) | 0 (0)
DUODENAL ULCER (Gastrointestinal disorders) | 1 (2) | 0 (0)
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 3 (3) | 0 (0)
GASTROINTESTINAL POLYP HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ILEAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
ILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ILEUS PARALYTIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 4 (4) | 0 (0)
INGUINAL HERNIA STRANGULATED (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 2 (2) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL POLYP (Gastrointestinal disorders) | 2 (2) | 0 (0)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 2 (2) | 0 (0)
MELAENA (Gastrointestinal disorders) | 1 (1) | 0 (0)
MESENTERIC ARTERY STENOSIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
OESOPHAGEAL RUPTURE (Gastrointestinal disorders) | 0 (0) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 3 (3) | 0 (0)
PERIODONTAL INFLAMMATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
PERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
RETROPERITONEAL HAEMATOMA (Gastrointestinal disorders) | 1 (1) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ADVERSE DRUG REACTION (General disorders) | 2 (2) | 0 (0)
CALCINOSIS (General disorders) | 1 (1) | 0 (0)
CATHETER SITE HAEMATOMA (General disorders) | 1 (1) | 0 (0)
CHEST PAIN (Gastrointestinal disorders) | 6 (6) | 0 (0)
DEATH (General disorders) | 6 (6) | 0 (0)
DEVICE BATTERY ISSUE (General disorders) | 1 (1) | 0 (0)
DEVICE MALFUNCTION (General disorders) | 1 (1) | 0 (0)
DEVICE OCCLUSION (Gastrointestinal disorders) | 13 (14) | 7 (9)
GENERAL PHYSICAL HEALTH DETERIORATION (Gastrointestinal disorders) | 3 (4) | 1 (1)
HERNIA (General disorders) | 0 (0) | 1 (1)
IMPAIRED HEALING (General disorders) | 2 (2) | 1 (1)
IMPAIRED SELF-CARE (General disorders) | 1 (1) | 0 (0)
INJECTION SITE HAEMORRHAGE (General disorders) | 1 (1) | 0 (0)
MALAISE (General disorders) | 1 (1) | 0 (0)
OBSTRUCTION (General disorders) | 1 (1) | 0 (0)
PAIN (General disorders) | 3 (3) | 0 (0)
POLYP (General disorders) | 1 (1) | 0 (0)
PUNCTURE SITE HAEMORRHAGE (General disorders) | 2 (2) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 1 (1)
STENT-GRAFT ENDOLEAK (General disorders) | 1 (2) | 0 (0)
STENT MALFUNCTION (General disorders) | 0 (0) | 2 (2)
SUDDEN DEATH (General disorders) | 1 (1) | 0 (0)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 1 (1) | 0 (0)
BILIARY COLIC (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLANGITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 5 (5) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC LESION (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
CONTRAST MEDIA ALLERGY (Immune system disorders) | 2 (2) | 0 (0)
ABDOMINAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
ABSCESS LIMB (Infections and infestations) | 1 (1) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 1 (1) | 0 (0)
ARTHRITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
BACTERAEMIA (Infections and infestations) | 2 (2) | 0 (0)
BACTERIAL INFECTION (Infections and infestations) | 2 (2) | 0 (0)
BLISTER INFECTED (Infections and infestations) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 6 (6) | 1 (1)
BRONCHOPNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
CANDIDA INFECTION (Infections and infestations) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 3 (3) | 0 (0)
CORONA VIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
CYSTITIS (Infections and infestations) | 1 (1) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1) | 0 (0)
DEVICE RELATED SEPSIS (Infections and infestations) | 1 (2) | 0 (0)
ENDOCARDITIS (Infections and infestations) | 3 (3) | 0 (0)
ERYSIPELAS (Infections and infestations) | 1 (1) | 0 (0)
GANGRENE (Infections and infestations) | 3 (3) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0)
GROIN INFECTION (Infections and infestations) | 2 (2) | 0 (0)
ILEAL GANGRENE (Infections and infestations) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 5 (5) | 0 (0)
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 1 (1) | 1 (1)
INFLUENZA (Infections and infestations) | 2 (2) | 0 (0)
LIVER ABSCESS (Infections and infestations) | 1 (2) | 0 (0)
LOCALISED INFECTION (Infections and infestations) | 3 (3) | 0 (0)
LUNG INFECTION (Infections and infestations) | 2 (2) | 0 (0)
MEDIASTINAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
MYCOTIC ANEURYSM (Infections and infestations) | 1 (1) | 0 (0)
ORCHITIS (Infections and infestations) | 1 (1) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 4 (4) | 0 (0)
PELVIC ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
PERITONITIS (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 19 (24) | 4 (4)
PSOAS ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
PULPITIS DENTAL (Infections and infestations) | 1 (1) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 1 (1) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 5 (5) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 2 (2) | 0 (0)
SINUSITIS (Infections and infestations) | 1 (1) | 0 (0)
SOFT TISSUE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 5 (5) | 0 (0)
UROSEPSIS (Infections and infestations) | 3 (3) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 3 (3) | 0 (0)
WOUND INFECTION (Infections and infestations) | 2 (2) | 0 (0)
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ARTERIAL RESTENOSIS (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
CRANIOCEREBRAL INJURY (Infections and infestations) | 1 (1) | 0 (0)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 5 (6) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
GRAFT THROMBOSIS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
INJURY (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
KIDNEY CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LIMB INJURY (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
MENISCUS INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
PERIPHERAL ARTERIAL REOCCLUSION (Injury, poisoning and procedural complications) | 11 (17) | 1 (1)
PERIPHERAL ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 39 (54) | 6 (6)
POST PROCEDURAL FISTULA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POSTOPERATIVE WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PUBIS FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
REOCCLUSION (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
SEROMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SOFT TISSUE INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
SPLENIC RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
TENDON INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
TOOTH INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
TRACHEAL INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
VASCULAR GRAFT OCCLUSION (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 8 (8) | 1 (1)
WOUND (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
WOUND EVISCERATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WOUND HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
ANGIOGRAM (Investigations) | 2 (2) | 1 (1)
ANGIOGRAM PERIPHERAL (Investigations) | 1 (1) | 0 (0)
BLOOD URINE PRESENT (Investigations) | 1 (1) | 0 (0)
BORDETELLA TEST POSITIVE (Investigations) | 1 (1) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 1 (1) | 0 (0)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 1 (1) | 0 (0)
INVESTIGATION (Investigations) | 1 (1) | 0 (0)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 1 (1)
LYMPH NODES SCAN ABNORMAL (Investigations) | 0 (0) | 1 (1)
CACHEXIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OBESITY (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (3)
BURSITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
COMPARTMENT SYNDROME (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 9 (9) | 0 (0)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
PLANTAR FASCIAL FIBROMATOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
POLYMYALGIA RHEUMATICA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ANOGENITAL WARTS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
BREAST CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CARCINOID TUMOUR OF THE GASTROINTESTINAL TRACT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CHOLANGIOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
COLON CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COLORECTAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
EAR NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
GLIOBLASTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
HEPATIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
HODGKIN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
LUNG ADENOCARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG CARCINOMA CELL TYPE UNSPECIFIED RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 0 (0)
LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MAXILLOFACIAL SINUS NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
OESOPHAGEAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OROPHARYNGEAL SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PLASMA CELL MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
PROSTATE CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PROSTATIC ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SALIVARY GLAND CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
TUMOUR OF AMPULLA OF VATER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
URETHRAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
VULVAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 5 (5) | 2 (2)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 1 (1) | 1 (2)
CEREBRAL ARTERY OCCLUSION (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 8 (8) | 1 (1)
DEMENTIA (Nervous system disorders) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1)
FACIAL SPASM (Nervous system disorders) | 1 (1) | 0 (0)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 (1) | 0 (0)
ISCHAEMIC CEREBRAL INFARCTION (Nervous system disorders) | 1 (1) | 0 (0)
LACUNAR INFARCTION (Nervous system disorders) | 2 (2) | 0 (0)
MOTOR NEURONE DISEASE (Nervous system disorders) | 1 (1) | 0 (0)
NORMAL PRESSURE HYDROCEPHALUS (Nervous system disorders) | 1 (2) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 2 (2) | 0 (0)
PARKINSON'S DISEASE (Nervous system disorders) | 1 (1) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 3 (3) | 0 (0)
RADICULOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 8 (8) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 7 (8) | 0 (0)
VIITH NERVE PARALYSIS (Nervous system disorders) | 1 (1) | 0 (0)
AGGRESSION (Psychiatric disorders) | 0 (0) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 0 (0)
DELIRIUM (Psychiatric disorders) | 2 (2) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0)
MENTAL DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 1 (1)
BLADDER PERFORATION (Renal and urinary disorders) | 1 (1) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 3 (5) | 1 (1)
HAEMORRHAGE URINARY TRACT (Renal and urinary disorders) | 1 (1) | 0 (0)
MICTURITION DISORDER (Renal and urinary disorders) | 1 (1) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 2 (2) | 1 (1)
NOCTURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 2 (2) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 12 (12) | 1 (1)
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL IMPAIRMENT (Renal and urinary disorders) | 3 (3) | 0 (0)
URETHRAL DILATATION (Renal and urinary disorders) | 1 (1) | 0 (0)
URETHRAL MEATUS STENOSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
URETHRAL STENOSIS (Renal and urinary disorders) | 1 (2) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 3 (3) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 4 (4) | 0 (0)
PROSTATIC HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
PROSTATITIS (Reproductive system and breast disorders) | 1 (1) | 0 (0)
VAGINAL PROLAPSE (Reproductive system and breast disorders) | 2 (2) | 0 (0)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
BRONCHIAL DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
NASAL SEPTUM DEVIATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PNEUMOTHORAX SPONTANEOUS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 0 (0)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATOMYOSITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DIABETIC FOOT (Skin and subcutaneous tissue disorders) | 4 (7) | 0 (0)
PETECHIAE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PSORIASIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 6 (7) | 1 (1)
ANGIOPLASTY (Surgical and medical procedures) | 1 (1) | 0 (0)
ALCOHOL DETOXIFICATION (Surgical and medical procedures) | 0 (0) | 1 (1)
CARDIAC OPERATION (Surgical and medical procedures) | 1 (1) | 0 (0)
DEBRIDEMENT (Surgical and medical procedures) | 1 (1) | 0 (0)
DUPUYTREN'S CONTRACTURE OPERATION (Surgical and medical procedures) | 1 (1) | 0 (0)
EYE OPERATION (Surgical and medical procedures) | 1 (1) | 0 (0)
GASTROSTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
HIP ARTHROPLASTY (Surgical and medical procedures) | 1 (1) | 0 (0)
HIP SURGERY (Surgical and medical procedures) | 2 (2) | 0 (0)
ILEOSTOMY CLOSURE (Surgical and medical procedures) | 1 (1) | 0 (0)
INTESTINAL RESECTION (Surgical and medical procedures) | 1 (1) | 0 (0)
KNEE OPERATION (Surgical and medical procedures) | 2 (2) | 0 (0)
LEG AMPUTATION (Surgical and medical procedures) | 1 (1) | 0 (0)
LIVER ABLATION (Surgical and medical procedures) | 1 (1) | 0 (0)
MEDICAL DEVICE CHANGE (Surgical and medical procedures) | 1 (1) | 0 (0)
NASAL CYST REMOVAL (Surgical and medical procedures) | 1 (1) | 0 (0)
OESOPHAGECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
PERIPHERAL ARTERY ANGIOPLASTY (Surgical and medical procedures) | 1 (1) | 0 (0)
PERIPHERAL ARTERY BYPASS (Surgical and medical procedures) | 1 (1) | 0 (0)
PERIPHERAL REVASCULARISATION (Surgical and medical procedures) | 4 (6) | 0 (0)
RADICAL PROSTATECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
SKIN NEOPLASM EXCISION (Surgical and medical procedures) | 1 (3) | 0 (0)
SPINAL LAMINECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
TENDON OPERATION (Surgical and medical procedures) | 0 (0) | 1 (1)
THROMBECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
THROMBOLYSIS (Surgical and medical procedures) | 1 (1) | 0 (0)
THYROID OPERATION (Surgical and medical procedures) | 1 (1) | 0 (0)
AORTIC ANEURYSM (Vascular disorders) | 2 (2) | 0 (0)
AORTIC STENOSIS (Vascular disorders) | 3 (3) | 0 (0)
ARTERIAL DISORDER (Vascular disorders) | 1 (1) | 0 (0)
ARTERIAL HAEMORRHAGE (Vascular disorders) | 2 (2) | 0 (0)
ARTERIAL SPASM (Vascular disorders) | 1 (1) | 0 (0)
ARTERIAL STENOSIS (Vascular disorders) | 4 (4) | 1 (1)
ARTERIOSCLEROSIS (Vascular disorders) | 1 (1) | 1 (1)
ARTERIOVENOUS FISTULA (Vascular disorders) | 1 (1) | 0 (0)
EXTREMITY NECROSIS (Vascular disorders) | 1 (2) | 0 (0)
FEMORAL ARTERY DISSECTION (Vascular disorders) | 32 (32) | 0 (0)
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 27 (33) | 4 (4)
FLUSHING (Vascular disorders) | 1 (1) | 0 (0)
HAEMATOMA (Vascular disorders) | 3 (3) | 1 (1)
HAEMODYNAMIC INSTABILITY (Vascular disorders) | 1 (1) | 0 (0)
HAEMORRHAGE (Vascular disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0)
HYPERTENSIVE CRISIS (Vascular disorders) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 1 (1)
HYPOVOLAEMIC SHOCK (Vascular disorders) | 1 (1) | 0 (0)
ILIAC ARTERY OCCLUSION (Vascular disorders) | 1 (1) | 0 (0)
INTERMITTENT CLAUDICATION (Vascular disorders) | 34 (44) | 6 (7)
MACROANGIOPATHY (Vascular disorders) | 1 (1) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 16 (18) | 1 (1)
PERIPHERAL ARTERY ANEURYSM (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL ARTERY DISSECTION (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 91 (132) | 16 (23)
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 4 (4) | 0 (0)
PERIPHERAL EMBOLISM (Vascular disorders) | 6 (6) | 1 (1)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 8 (8) | 1 (1)
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 4 (6) | 0 (0)
TEMPORAL ARTERITIS (Vascular disorders) | 1 (1) | 0 (0)
VARICOSE VEIN (Vascular disorders) | 1 (1) | 0 (0)
VASCULAR CALCIFICATION (Vascular disorders) | 1 (1) | 0 (0)
VASOSPASM (Vascular disorders) | 4 (4) | 0 (0)
VESSEL PERFORATION (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Global Cohort 1 (N=370) | Global ISR Cohort 2 (N=122)
CATHETER SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 17 (18) | 0 (0)
AUTOIMMUNE HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
HAEMORRHAGIC DISORDER (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
IMMUNE THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
NORMOCHROMIC NORMOCYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
THROMBOCYTOSIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 (1) | 0 (0)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 2 (2) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 18 (19) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 16 (19) | 1 (1)
ANGINA UNSTABLE (Cardiac disorders) | 7 (9) | 0 (0)
AORTIC VALVE STENOSIS (Cardiac disorders) | 5 (6) | 0 (0)
ARRHYTHMIA (Cardiac disorders) | 1 (2) | 0 (0)
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 24 (27) | 1 (1)
ATRIAL FLUTTER (Cardiac disorders) | 5 (17) | 0 (0)
BRADYARRHYTHMIA (Cardiac disorders) | 1 (1) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 2 (2) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 2 (2) | 0 (0)
CARDIAC DISORDER (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 11 (18) | 2 (2)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 6 (12) | 0 (0)
CARDIAC SEPTAL HYPERTROPHY (Cardiac disorders) | 1 (1) | 0 (0)
CARDIOGENIC SHOCK (Cardiac disorders) | 1 (1) | 0 (0)
CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1)
COR PULMONALE ACUTE (Cardiac disorders) | 1 (1) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 17 (21) | 4 (4)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 3 (4) | 0 (0)
DIASTOLIC DYSFUNCTION (Cardiac disorders) | 1 (1) | 0 (0)
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 4 (4) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 4 (4) | 1 (1)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 3 (3) | 0 (0)
PALPITATIONS (Cardiac disorders) | 3 (4) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1) | 0 (0)
PRINZMETAL ANGINA (Cardiac disorders) | 1 (1) | 0 (0)
SICK SINUS SYNDROME (Cardiac disorders) | 1 (1) | 0 (0)
STRESS CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 0 (0)
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 2 (2) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 3 (3) | 0 (0)
TACHYARRHYTHMIA (Cardiac disorders) | 2 (2) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 6 (6) | 0 (0)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 2 (2) | 0 (0)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 3 (3) | 0 (0)
HAMARTOMA (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
HYDROCELE (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
DEAFNESS (Ear and labyrinth disorders) | 1 (1) | 0 (0)
MENIERE'S DISEASE (Ear and labyrinth disorders) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 3 (4) | 4 (4)
GOITRE (Endocrine disorders) | 1 (1) | 0 (0)
HYPERPARATHYROIDISM (Endocrine disorders) | 2 (2) | 0 (0)
HYPERTHYROIDISM (Endocrine disorders) | 3 (3) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1) | 1 (1)
THYROID CYST (Endocrine disorders) | 1 (1) | 0 (0)
AMAUROSIS FUGAX (Eye disorders) | 1 (1) | 0 (0)
CATARACT (Eye disorders) | 5 (6) | 0 (0)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 1 (1) | 0 (0)
CORNEAL DECOMPENSATION (Eye disorders) | 1 (1) | 0 (0)
DIABETIC RETINOPATHY (Eye disorders) | 0 (0) | 1 (2)
ECTROPION (Eye disorders) | 1 (1) | 0 (0)
ENTROPION (Eye disorders) | 1 (1) | 0 (0)
EYE HAEMORRHAGE (Eye disorders) | 1 (1) | 0 (0)
EYELID PTOSIS (Eye disorders) | 0 (0) | 1 (1)
LAGOPHTHALMOS (Eye disorders) | 1 (1) | 0 (0)
MACULAR FIBROSIS (Eye disorders) | 2 (2) | 0 (0)
RETINAL VEIN OCCLUSION (Eye disorders) | 2 (2) | 0 (0)
RETINOPATHY (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 (1) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 (9) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0)
BARRETT'S OESOPHAGUS (Gastrointestinal disorders) | 2 (3) | 1 (1)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 0 (0)
DENTAL CARIES (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIAPHRAGMATIC HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 6 (7) | 0 (0)
DIVERTICULITIS INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIVERTICULUM (Gastrointestinal disorders) | 2 (2) | 0 (0)
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 1 (1) | 0 (0)
DUODENAL ULCER (Gastrointestinal disorders) | 1 (2) | 0 (0)
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 4 (4) | 0 (0)
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC POLYPS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 5 (6) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 3 (3) | 0 (0)
GASTROINTESTINAL POLYP HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2) | 0 (0)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 1 (1)
HAEMORRHOIDS THROMBOSED (Gastrointestinal disorders) | 1 (1) | 0 (0)
ILEAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
ILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ILEUS PARALYTIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 6 (6) | 0 (0)
INGUINAL HERNIA STRANGULATED (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 2 (2) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL POLYP (Gastrointestinal disorders) | 3 (3) | 0 (0)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 3 (3) | 0 (0)
MELAENA (Gastrointestinal disorders) | 4 (4) | 0 (0)
MESENTERIC ARTERY STENOSIS (Gastrointestinal disorders) | 3 (3) | 0 (0)
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 3 (3) | 0 (0)
OESOPHAGEAL RUPTURE (Gastrointestinal disorders) | 0 (0) | 1 (1)
OESOPHAGITIS (Gastrointestinal disorders) | 1 (2) | 0 (0)
PANCREATIC CYST (Gastrointestinal disorders) | 1 (1) | 0 (0)
PANCREATIC MASS (Gastrointestinal disorders) | 1 (1) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 3 (3) | 0 (0)
PERIODONTAL INFLAMMATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
PERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
RETROPERITONEAL HAEMATOMA (Gastrointestinal disorders) | 1 (1) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 1 (1)
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ADVERSE DRUG REACTION (General disorders) | 3 (4) | 0 (0)
ASTHENIA (General disorders) | 1 (1) | 0 (0)
CALCINOSIS (General disorders) | 1 (1) | 0 (0)
CATHETER SITE BRUISE (General disorders) | 4 (5) | 0 (0)
CATHETER SITE DISCHARGE (General disorders) | 7 (7) | 0 (0)
CATHETER SITE HAEMATOMA (General disorders) | 5 (5) | 1 (1)
CATHETER SITE HAEMORRHAGE (General disorders) | 7 (7) | 1 (1)
CATHETER SITE RELATED REACTION (General disorders) | 1 (1) | 0 (0)
CHEST DISCOMFORT (General disorders) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 13 (13) | 3 (3)
CYST (General disorders) | 1 (1) | 1 (1)
DEATH (General disorders) | 6 (6) | 0 (0)
DEVICE BATTERY ISSUE (General disorders) | 1 (1) | 0 (0)
DEVICE MALFUNCTION (General disorders) | 1 (1) | 0 (0)
DEVICE OCCLUSION (General disorders) | 15 (18) | 9 (11)
DISCOMFORT (General disorders) | 1 (1) | 0 (0)
DRUG INTOLERANCE (General disorders) | 1 (1) | 0 (0)
EFFUSION (General disorders) | 1 (1) | 0 (0)
EXERCISE TOLERANCE DECREASED (General disorders) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 1 (1) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 3 (4) | 1 (1)
HERNIA (General disorders) | 0 (0) | 1 (1)
IMPAIRED HEALING (General disorders) | 4 (4) | 1 (1)
IMPAIRED SELF-CARE (General disorders) | 1 (1) | 0 (0)
INJECTION SITE HAEMORRHAGE (General disorders) | 1 (1) | 0 (0)
LOCAL SWELLING (General disorders) | 9 (9) | 1 (1)
MALAISE (General disorders) | 1 (1) | 0 (0)
OBSTRUCTION (General disorders) | 1 (1) | 0 (0)
OEDEMA (General disorders) | 3 (3) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 9 (9) | 0 (0)
PAIN (General disorders) | 5 (5) | 2 (2)
POLYP (General disorders) | 1 (2) | 0 (0)
PUNCTURE SITE DISCHARGE (General disorders) | 2 (2) | 0 (0)
PUNCTURE SITE HAEMORRHAGE (General disorders) | 4 (5) | 2 (2)
PUNCTURE SITE PAIN (General disorders) | 4 (5) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 1 (1)
STENT-GRAFT ENDOLEAK (General disorders) | 1 (2) | 0 (0)
STENT MALFUNCTION (General disorders) | 0 (0) | 2 (2)
SUDDEN DEATH (General disorders) | 1 (1) | 0 (0)
SWELLING (General disorders) | 0 (0) | 1 (1)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 1 (1) | 0 (0)
THROMBOSIS IN DEVICE (General disorders) | 0 (0) | 1 (1)
VESSEL PUNCTURE SITE DISCHARGE (General disorders) | 1 (1) | 0 (0)
VESSEL PUNCTURE SITE HAEMATOMA (General disorders) | 1 (1) | 0 (0)
BILIARY COLIC (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLANGITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 6 (6) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 3 (3) | 0 (0)
HEPATIC ARTERY STENOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC LESION (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
CONTRAST MEDIA ALLERGY (Immune system disorders) | 2 (2) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 0 (0)
ABDOMINAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
ABSCESS LIMB (Infections and infestations) | 1 (1) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 2 (2) | 0 (0)
APPENDICITIS (Infections and infestations) | 1 (1) | 0 (0)
ARTHRITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
BACTERAEMIA (Infections and infestations) | 2 (2) | 0 (0)
BACTERIAL INFECTION (Infections and infestations) | 2 (2) | 0 (0)
BACTERIURIA (Infections and infestations) | 1 (1) | 0 (0)
BLISTER INFECTED (Infections and infestations) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 8 (8) | 2 (2)
BRONCHOPNEUMONIA (Infections and infestations) | 1 (1) | 1 (1)
CANDIDA INFECTION (Infections and infestations) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 3 (6) | 0 (0)
CORONA VIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
CYSTITIS (Infections and infestations) | 2 (3) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1) | 0 (0)
DEVICE RELATED SEPSIS (Infections and infestations) | 1 (2) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 0 (0)
EAR INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ENDOCARDITIS (Infections and infestations) | 3 (3) | 0 (0)
ENTEROCOCCAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ERYSIPELAS (Infections and infestations) | 2 (2) | 0 (0)
FURUNCLE (Infections and infestations) | 2 (2) | 0 (0)
GANGRENE (Infections and infestations) | 3 (3) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS NOROVIRUS (Infections and infestations) | 1 (1) | 0 (0)
GROIN INFECTION (Infections and infestations) | 2 (2) | 0 (0)
HELICOBACTER INFECTION (Infections and infestations) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 2 (2) | 0 (0)
ILEAL GANGRENE (Infections and infestations) | 1 (1) | 0 (0)
INFECTED BITES (Infections and infestations) | 1 (1) | 0 (0)
INFECTED DERMAL CYST (Infections and infestations) | 1 (1) | 0 (0)
INFECTED LYMPHOCELE (Infections and infestations) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 6 (6) | 0 (0)
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 1 (1) | 1 (1)
INFLUENZA (Infections and infestations) | 7 (7) | 0 (0)
LIVER ABSCESS (Infections and infestations) | 1 (2) | 0 (0)
LOCALISED INFECTION (Infections and infestations) | 3 (3) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0)
LUNG INFECTION (Infections and infestations) | 2 (2) | 0 (0)
MEDIASTINAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
MYCOTIC ANEURYSM (Infections and infestations) | 1 (1) | 0 (0)
NAIL BED INFECTION (Infections and infestations) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 7 (7) | 2 (2)
OPHTHALMIC HERPES ZOSTER (Infections and infestations) | 1 (1) | 0 (0)
ORCHITIS (Infections and infestations) | 2 (2) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 5 (5) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 1 (1) | 0 (0)
PELVIC ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
PERITONITIS (Infections and infestations) | 1 (1) | 0 (0)
PHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 21 (27) | 4 (4)
PSOAS ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
PULPITIS DENTAL (Infections and infestations) | 2 (2) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 1 (1) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0)
SEPSIS (Infections and infestations) | 5 (5) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 2 (2) | 0 (0)
SIALOADENITIS (Infections and infestations) | 1 (1) | 0 (0)
SINUSITIS (Infections and infestations) | 3 (3) | 0 (0)
SKIN INFECTION (Infections and infestations) | 1 (1) | 0 (0)
SOFT TISSUE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (6) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 12 (13) | 2 (2)
UROSEPSIS (Infections and infestations) | 3 (3) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 4 (5) | 0 (0)
WOUND INFECTION (Infections and infestations) | 3 (5) | 0 (0)
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ARTERIAL RESTENOSIS (Injury, poisoning and procedural complications) | 3 (3) | 7 (7)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
BREAST INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
BURNS THIRD DEGREE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CAROTID ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CONCUSSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 9 (11) | 2 (2)
CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 10 (13) | 1 (1)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
GRAFT THROMBOSIS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HAND FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
INFLAMMATION OF WOUND (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INJURY (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
JOINT INJURY (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
KIDNEY CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
LIMB INJURY (Injury, poisoning and procedural complications) | 7 (8) | 0 (0)
MENISCUS INJURY (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
NAIL INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
PERIORBITAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PERIPHERAL ARTERIAL REOCCLUSION (Injury, poisoning and procedural complications) | 13 (24) | 1 (3)
PERIPHERAL ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 70 (103) | 10 (13)
POST PROCEDURAL FISTULA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL SWELLING (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POSTOPERATIVE ILEUS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POSTOPERATIVE WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PROCEDURAL HEADACHE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
PROCEDURAL HYPERTENSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PUBIS FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
REOCCLUSION (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
SCAPULA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SEROMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SKIN WOUND (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SOFT TISSUE INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
SPLENIC RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TENDON INJURY (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
TOOTH INJURY (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
TRACHEAL INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
URINARY RETENTION POSTOPERATIVE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
VASCULAR GRAFT OCCLUSION (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 9 (9) | 2 (2)
WOUND (Injury, poisoning and procedural complications) | 6 (6) | 6 (7)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 3 (4) | 0 (0)
WOUND EVISCERATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WOUND HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
WOUND NECROSIS (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
ANGIOGRAM (Investigations) | 2 (2) | 1 (1)
ANGIOGRAM PERIPHERAL (Investigations) | 1 (1) | 0 (0)
ANKLE BRACHIAL INDEX DECREASED (Investigations) | 4 (4) | 0 (0)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 3 (3) | 1 (1)
BLOOD GLUCOSE ABNORMAL (Investigations) | 1 (2) | 0 (0)
BLOOD URINE PRESENT (Investigations) | 1 (1) | 0 (0)
BODY TEMPERATURE DECREASED (Investigations) | 1 (1) | 0 (0)
BORDETELLA TEST POSITIVE (Investigations) | 1 (1) | 0 (0)
C-REACTIVE PROTEIN INCREASED (Investigations) | 1 (1) | 0 (0)
CARDIAC MURMUR (Investigations) | 1 (1) | 0 (0)
COMA SCALE (Investigations) | 1 (1) | 0 (0)
ELECTROCARDIOGRAM ST SEGMENT ELEVATION (Investigations) | 2 (2) | 0 (0)
ENDOSCOPY UPPER GASTROINTESTINAL TRACT (Investigations) | 1 (1) | 0 (0)
GLYCOSYLATED HAEMOGLOBIN INCREASED (Investigations) | 1 (1) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 2 (2) | 0 (0)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 1 (1) | 0 (0)
INVESTIGATION (Investigations) | 1 (1) | 0 (0)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 1 (1)
LYMPH NODES SCAN ABNORMAL (Investigations) | 0 (0) | 2 (2)
PROSTATIC SPECIFIC ANTIGEN INCREASED (Investigations) | 1 (1) | 0 (0)
RED BLOOD CELL COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
CACHEXIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
GOUT (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 (5) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 5 (6) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
IRON DEFICIENCY (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
MALNUTRITION (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
OBESITY (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
VITAMIN B12 DEFICIENCY (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 15 (16) | 4 (4)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 21 (22) | 8 (10)
BURSITIS (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
COMPARTMENT SYNDROME (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
EXOSTOSIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
GOUTY ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LIMB DISCOMFORT (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
MUSCLE ATROPHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 14 (14) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 7 (7) | 0 (0)
MYOSCLEROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OSTEITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 18 (21) | 2 (2)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 43 (49) | 7 (11)
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PLANTAR FASCIAL FIBROMATOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PLANTAR FASCIITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
POLYMYALGIA RHEUMATICA (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
SCOLIOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SENSATION OF HEAVINESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ADRENAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ANOGENITAL WARTS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5) | 0 (0)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
BREAST CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CARCINOID TUMOUR OF THE GASTROINTESTINAL TRACT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CHOLANGIOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
COLON CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COLORECTAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
EAR NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
GLIOBLASTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
HAEMANGIOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
HAEMANGIOMA OF LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
HEPATIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
HODGKIN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
KERATOACANTHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LARYNGEAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LIPOMA OF BREAST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
LUNG ADENOCARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG CARCINOMA CELL TYPE UNSPECIFIED RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 0 (0)
LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
MAXILLOFACIAL SINUS NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
OESOPHAGEAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OROPHARYNGEAL SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PANCREATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PLASMA CELL MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 0 (0)
PROSTATE CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PROSTATIC ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SALIVARY GLAND CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
TUMOUR OF AMPULLA OF VATER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
URETHRAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
VULVAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BALANCE DISORDER (Nervous system disorders) | 1 (1) | 0 (0)
BURNING SENSATION (Nervous system disorders) | 2 (2) | 0 (0)
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 2 (2) | 0 (0)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 9 (13) | 3 (5)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 3 (5) | 1 (2)
CEREBRAL ARTERY OCCLUSION (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL HAEMATOMA (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 8 (8) | 1 (1)
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 1 (1) | 0 (0)
COGNITIVE DISORDER (Nervous system disorders) | 1 (1) | 0 (0)
DEMENTIA (Nervous system disorders) | 2 (2) | 0 (0)
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 2 (2) | 0 (0)
DIZZINESS (Nervous system disorders) | 3 (3) | 3 (3)
DYSAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0)
EPILEPSY (Nervous system disorders) | 1 (1) | 0 (0)
FACIAL SPASM (Nervous system disorders) | 1 (1) | 0 (0)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 3 (3) | 0 (0)
HEMIPLEGIA (Nervous system disorders) | 1 (1) | 0 (0)
HYPOTONIA (Nervous system disorders) | 0 (0) | 1 (1)
ISCHAEMIC CEREBRAL INFARCTION (Nervous system disorders) | 1 (1) | 0 (0)
LACUNAR INFARCTION (Nervous system disorders) | 2 (2) | 0 (0)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 0 (0)
MOTOR NEURONE DISEASE (Nervous system disorders) | 1 (1) | 0 (0)
NEURALGIA (Nervous system disorders) | 0 (0) | 1 (1)
NEURITIS (Nervous system disorders) | 1 (1) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 2 (2) | 0 (0)
NORMAL PRESSURE HYDROCEPHALUS (Nervous system disorders) | 1 (2) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 5 (5) | 1 (1)
PARKINSON'S DISEASE (Nervous system disorders) | 1 (1) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)
PERONEAL NERVE PALSY (Nervous system disorders) | 1 (1) | 0 (0)
PHANTOM PAIN (Nervous system disorders) | 1 (1) | 0 (0)
POLYNEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 4 (4) | 1 (1)
RADICULITIS LUMBOSACRAL (Nervous system disorders) | 1 (1) | 0 (0)
RADICULOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
RESTLESS LEGS SYNDROME (Nervous system disorders) | 1 (1) | 0 (0)
SCIATICA (Nervous system disorders) | 2 (2) | 1 (1)
SENSORY LOSS (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 11 (13) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 9 (10) | 0 (0)
TREMOR (Nervous system disorders) | 1 (1) | 0 (0)
VASCULAR DEMENTIA (Nervous system disorders) | 1 (1) | 0 (0)
VIITH NERVE PARALYSIS (Nervous system disorders) | 2 (2) | 0 (0)
AGGRESSION (Psychiatric disorders) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (2) | 0 (0)
BREATHING-RELATED SLEEP DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 0 (0)
DELIRIUM (Psychiatric disorders) | 3 (3) | 1 (1)
DEPRESSION (Psychiatric disorders) | 2 (3) | 0 (0)
EMOTIONAL DISTRESS (Psychiatric disorders) | 1 (1) | 0 (0)
MENTAL DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
POST-TRAUMATIC STRESS DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 1 (1)
BLADDER PERFORATION (Renal and urinary disorders) | 1 (1) | 0 (0)
CALCULUS BLADDER (Renal and urinary disorders) | 1 (1) | 0 (0)
CALCULUS URINARY (Renal and urinary disorders) | 2 (2) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 8 (11) | 1 (1)
HAEMORRHAGE URINARY TRACT (Renal and urinary disorders) | 1 (1) | 0 (0)
KIDNEY ENLARGEMENT (Renal and urinary disorders) | 1 (1) | 0 (0)
MICTURITION DISORDER (Renal and urinary disorders) | 1 (2) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 3 (3) | 1 (1)
NEPHROPATHY (Renal and urinary disorders) | 0 (0) | 1 (1)
NOCTURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
PRERENAL FAILURE (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 4 (4) | 0 (0)
RENAL CYST (Renal and urinary disorders) | 1 (1) | 2 (2)
RENAL FAILURE (Renal and urinary disorders) | 8 (8) | 2 (2)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 15 (16) | 1 (1)
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 7 (8) | 0 (0)
RENAL HYPERTENSION (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL IMPAIRMENT (Renal and urinary disorders) | 4 (4) | 0 (0)
URETHRAL DILATATION (Renal and urinary disorders) | 1 (1) | 0 (0)
URETHRAL MEATUS STENOSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
URETHRAL STENOSIS (Renal and urinary disorders) | 1 (2) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 2 (2) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 4 (4) | 0 (0)
ATROPHIC VULVOVAGINITIS (Reproductive system and breast disorders) | 1 (1) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 5 (5) | 0 (0)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PROSTATIC HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
PROSTATISM (Reproductive system and breast disorders) | 1 (1) | 0 (0)
PROSTATITIS (Reproductive system and breast disorders) | 1 (1) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 2 (2) | 0 (0)
VAGINAL PROLAPSE (Reproductive system and breast disorders) | 3 (4) | 0 (0)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
BRONCHIAL DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 13 (17) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 1 (1)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPERVENTILATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPOVENTILATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
NASAL SEPTUM DEVIATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PNEUMOTHORAX SPONTANEOUS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 0 (0)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY VASCULAR DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
VOCAL CORD LEUKOPLAKIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COLD SWEAT (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
DERMAL CYST (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATOMYOSITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DIABETIC FOOT (Skin and subcutaneous tissue disorders) | 4 (9) | 0 (0)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
HYPERSENSITIVITY VASCULITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
INTERTRIGO (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PETECHIAE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PSORIASIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
SKIN HAEMORRHAGE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKIN LESION (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 7 (18) | 1 (1)
STASIS DERMATITIS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
SWELLING FACE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
ALCOHOL DETOXIFICATION (Surgical and medical procedures) | 0 (0) | 1 (1)
ANGIOPLASTY (Surgical and medical procedures) | 1 (1) | 0 (0)
CARDIAC OPERATION (Surgical and medical procedures) | 1 (1) | 0 (0)
DEBRIDEMENT (Surgical and medical procedures) | 1 (2) | 0 (0)
DUPUYTREN'S CONTRACTURE OPERATION (Surgical and medical procedures) | 1 (1) | 0 (0)
EYE OPERATION (Surgical and medical procedures) | 1 (1) | 0 (0)
GASTROSTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
HIP ARTHROPLASTY (Surgical and medical procedures) | 1 (1) | 0 (0)
HIP SURGERY (Surgical and medical procedures) | 2 (2) | 0 (0)
ILEOSTOMY CLOSURE (Surgical and medical procedures) | 1 (1) | 0 (0)
INTESTINAL RESECTION (Surgical and medical procedures) | 1 (1) | 0 (0)
KNEE OPERATION (Surgical and medical procedures) | 2 (2) | 0 (0)
LEG AMPUTATION (Surgical and medical procedures) | 1 (1) | 0 (0)
LIVER ABLATION (Surgical and medical procedures) | 1 (1) | 0 (0)
MEDICAL DEVICE CHANGE (Surgical and medical procedures) | 1 (1) | 0 (0)
NASAL CYST REMOVAL (Surgical and medical procedures) | 1 (1) | 0 (0)
NERVE BLOCK (Surgical and medical procedures) | 1 (1) | 0 (0)
OESOPHAGECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
PERIPHERAL ARTERY ANGIOPLASTY (Surgical and medical procedures) | 1 (1) | 0 (0)
PERIPHERAL ARTERY BYPASS (Surgical and medical procedures) | 1 (1) | 0 (0)
PERIPHERAL REVASCULARISATION (Surgical and medical procedures) | 5 (7) | 0 (0)
POLYPECTOMY (Surgical and medical procedures) | 0 (0) | 1 (1)
RADICAL PROSTATECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
SKIN NEOPLASM EXCISION (Surgical and medical procedures) | 1 (3) | 0 (0)
SPINAL LAMINECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
TENDON OPERATION (Surgical and medical procedures) | 0 (0) | 1 (1)
THROMBECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
THROMBOLYSIS (Surgical and medical procedures) | 1 (1) | 0 (0)
THYROID OPERATION (Surgical and medical procedures) | 1 (1) | 0 (0)
ANEURYSM (Vascular disorders) | 1 (1) | 0 (0)
AORTIC ANEURYSM (Vascular disorders) | 5 (5) | 0 (0)
AORTIC DILATATION (Vascular disorders) | 1 (1) | 0 (0)
AORTIC STENOSIS (Vascular disorders) | 4 (4) | 0 (0)
ARTERIAL DISORDER (Vascular disorders) | 1 (1) | 1 (1)
ARTERIAL HAEMORRHAGE (Vascular disorders) | 2 (2) | 0 (0)
ARTERIAL SPASM (Vascular disorders) | 2 (2) | 0 (0)
ARTERIAL STENOSIS (Vascular disorders) | 5 (6) | 5 (6)
ARTERIOSCLEROSIS (Vascular disorders) | 2 (2) | 1 (1)
ARTERIOVENOUS FISTULA (Vascular disorders) | 4 (4) | 0 (0)
ARTERY DISSECTION (Vascular disorders) | 0 (0) | 2 (2)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2) | 0 (0)
ENDOTHELIAL DYSFUNCTION (Vascular disorders) | 1 (1) | 0 (0)
EXTREMITY NECROSIS (Vascular disorders) | 2 (3) | 0 (0)
FEMORAL ARTERY ANEURYSM (Vascular disorders) | 1 (1) | 0 (0)
FEMORAL ARTERY DISSECTION (Vascular disorders) | 35 (36) | 1 (1)
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 40 (50) | 5 (6)
FIBROMUSCULAR DYSPLASIA (Vascular disorders) | 1 (1) | 0 (0)
FLUSHING (Vascular disorders) | 1 (1) | 0 (0)
HAEMATOMA (Vascular disorders) | 13 (14) | 4 (4)
HAEMODYNAMIC INSTABILITY (Vascular disorders) | 1 (1) | 0 (0)
HAEMORRHAGE (Vascular disorders) | 1 (1) | 0 (0)
HOT FLUSH (Vascular disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 12 (13) | 0 (0)
HYPERTENSIVE CRISIS (Vascular disorders) | 2 (2) | 1 (1)
HYPOTENSION (Vascular disorders) | 3 (3) | 1 (1)
HYPOVOLAEMIC SHOCK (Vascular disorders) | 1 (1) | 0 (0)
ILIAC ARTERY OCCLUSION (Vascular disorders) | 1 (3) | 0 (0)
INTERMITTENT CLAUDICATION (Vascular disorders) | 90 (127) | 14 (16)
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
LYMPHOEDEMA (Vascular disorders) | 1 (1) | 0 (0)
MACROANGIOPATHY (Vascular disorders) | 1 (1) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 2 (2) | 1 (1)
PENETRATING ATHEROSCLEROTIC ULCER (Vascular disorders) | 2 (2) | 0 (0)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 31 (39) | 2 (2)
PERIPHERAL ARTERY ANEURYSM (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL ARTERY DISSECTION (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 141 (260) | 25 (45)
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 4 (4) | 0 (0)
PERIPHERAL EMBOLISM (Vascular disorders) | 6 (6) | 1 (1)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 8 (8) | 1 (1)
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 6 (8) | 0 (0)
POOR PERIPHERAL CIRCULATION (Vascular disorders) | 0 (0) | 1 (1)
RAYNAUD'S PHENOMENON (Vascular disorders) | 1 (1) | 0 (0)
SUBCLAVIAN ARTERY STENOSIS (Vascular disorders) | 1 (1) | 0 (0)
TEMPORAL ARTERITIS (Vascular disorders) | 1 (1) | 0 (0)
THROMBOPHLEBITIS (Vascular disorders) | 2 (2) | 0 (0)
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 3 (3) | 0 (0)
THROMBOSIS (Vascular disorders) | 3 (3) | 0 (0)
VARICOSE VEIN (Vascular disorders) | 3 (3) | 0 (0)
VASCULAR CALCIFICATION (Vascular disorders) | 3 (4) | 0 (0)
VASCULAR RUPTURE (Vascular disorders) | 0 (0) | 1 (1)
VASOSPASM (Vascular disorders) | 4 (4) | 0 (0)
VENOUS HAEMORRHAGE (Vascular disorders) | 1 (1) | 0 (0)
VENOUS INSUFFICIENCY (Vascular disorders) | 2 (2) | 0 (0)
VESSEL PERFORATION (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-11-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT01927068/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/68/NCT01927068/SAP_001.pdf